CLINICAL TRIAL: NCT00866528
Title: An Open-label, Multicenter, Phase I/II Study of Pazopanib in Combination With Paclitaxel in First-line Treatment of Subjects With Stage IIIBwet/IV Non-small Cell Lung Cancer
Brief Title: Study of Pazopanib and Paclitaxel in Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111109
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: paclitaxel; NSCLC; pazopanib; Advanced Non-Small Cell Lung Cancer; non-small cell lung cancer; Advanced Solid Tumor; GW786034; Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase I (Experimental): oral pazopanib once daily (Phase I starting dose 800 mg) and paclitaxel IV once every 3 weeks (Phase I starting dose 135 mg/m2).
  Interventions: Drug: pazopanib; Drug: paclitaxel

INTERVENTIONS:
Drug: pazopanib — oral pazopanib once daily (Phase I starting dose 800 mg)
  Other Names: Votrient
Drug: paclitaxel — paclitaxel IV once every 3 weeks (Phase I starting dose 135 mg/m2).

SUMMARY:
The Phase I part of the study will identify the doses of pazopanib and paclitaxel that can be administered safely in combination. The Phase II part of the study will not be progressed as documented in Protocol Amendment 01.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* At least 18 years old
* Histologically- or cytologically-confirmed diagnosis of Stage IIIBwet (with confirmed malignant pleural effusion) or Stage IV NSCLC (or for Phase I only, advanced solid tumor for which there is no standard therapy or for whom paclitaxel is standard therapy).
* No prior systemic first-line therapy for advanced disease
* Measurable disease
* ECOG performance status of 0 or 1
* Life expectancy of at least 12 weeks.
* Able to swallow and retain oral medication
* Adequate organ system function (hematological, renal, and hepatic)
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) OR childbearing potential, and agrees to use adequate contraception

Exclusion Criteria:

* Active malignancy or any malignancy in the 3 years prior to first dose of study drug other than NSCLC (or for Phase I, other than the primary solid tumor)
* CNS metastases or leptomeningeal carcinomatosis, except for asymptomatic, previously treated CNS metastases
* Clinically significant gastrointestinal abnormalities
* Prolongation of corrected QT interval (QTc) > 480 msecs
* History of any one or more cardiovascular conditions within the past 6 months prior to randomization
* Poorly controlled hypertension
* History of cerebrovascular accident (including transient ischemic attacks), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Major surgery or trauma within 28 days or any non-healing wound, fracture, or ulcer
* Evidence of active bleeding or bleeding diathesis
* Recent hemoptysis
* Endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Serious and/or unstable pre-existing medical (e.g., uncontrolled infection), psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Use of any prohibited medication
* Use of an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug
* Ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity except alopecia
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib, paclitaxel, and/or carboplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07-09 (Actual); Primary Completion 2012-10-25 (Actual); Study Completion 2012-10-25 (Actual)

PRIMARY OUTCOMES:
Phase I: safety and tolerability (Serious adverse events, adverse events, dose-limiting toxicities, clinical laboratory data, vital signs, ECG, ECOG performance status) | at least one cycle of treatment (3 weeks)

SECONDARY OUTCOMES:
Phase I: paclitaxel and pazopanib pharmacokinetics | Cycle 1 and Cycle 2 PK sampling
Phase I: clinical activity | at least 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (2):
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Columbus, Ohio
- United Kingdom (2):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Newcastle upon Tyne

REFERENCES:
- See also: Results for study 111109 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111109?search=study&study_ids=111109#rs